CLINICAL TRIAL: NCT04152798
Title: Approach to Hiatal Hernia Repair Based on Collagen Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grubnik Volodymyr (Other)
Responsible Party: Sponsor-Investigator, Grubnik Volodymyr, MD, Professor, Odessa National Medical University
Organization: Odessa National Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONMedU
Record Dates: First submitted 2019-10-26; First posted 2019-11-05 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Hiatal Hernia; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

ARMS (2):
- ProGrip™ mesh repair (Active Comparator): Laparoscopic hiatal hernia repair with ProGrip™ mesh
  Interventions: Procedure: Laparoscopic hiatal hernia repair with ProGrip™ mesh
- Primary crural repair (Active Comparator): Primary posterior crura repair
  Interventions: Procedure: Laparoscopic primary posterior crural repair

INTERVENTIONS:
Procedure: Laparoscopic hiatal hernia repair with ProGrip™ mesh — Suturing of the right and left diaphragmatic crura using 3 to 4 interrupted nonabsorbable stitches with additional reinforcement of crura repair with ProGrip™ mesh
  Other Names: Laparoscopic mesh hiatoplasty; Laparoscopic mesh hiatal closure
  Arms: ProGrip™ mesh repair
Procedure: Laparoscopic primary posterior crural repair — Posterior cruroraphy will be performed with 3 to 4 interrupted non-absorbable sutures
  Other Names: Laparoscopic posterior crurorrhaphy; Laparoscopic posterior crural closure
  Arms: Primary crural repair

SUMMARY:
Groups of patients who underwent laparoscopic repair of large hiatal hernias by primary posterior crural repair and crural repair with ProGrip™ mesh techniques were examined for recurrence rate of hiatal hernias, quality of life according to the GERD-HRQL questionnaire. Clinical evaluation was performed at 3, 6, 12, 24, 36, and 48 months after surgery.

DETAILED DESCRIPTION:
The laparoscopic repair of large hiatal hernias is mostly performed by cruroraphy or cruroraphy with mesh reinforcement techniques.

Cruroraphy it is suturing of the right and left diaphragmatic crura using nonabsorbable stitches. Main disadvantage of such technique is the high hiatal hernia recurrence rate after surgery.

Cruroraphy with mesh reinforcement technique followed by relatively less hiatal hernia recurrence rate but associated with a large number of mesh-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 20 years
* Initially suffering from large hiatal hernia (>20% of the stomach in the thoracic cavity)
* Performance of laparoscopic hiatal hernia repair
* Informed Consent as documented by signature

Exclusion Criteria:

* Cases of conversion to open surgery
* Age < 20 years and > 80 years
* History of oesophageal/gastric/duodenal surgery including vagotomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of hiatal hernia | 36 months
  Recurrence of hiatal hernia will be assessed by barium contrast swallow study

SECONDARY OUTCOMES:
Quality of life and satisfaction | 36 months
  Quality of life and satisfaction will be assessed by Gastroesophageal reflux disease - health-related quality of life (GERD-HRQL) score. The scale has 11 items,each item is scored from 0 to 5. A higher score indicating a better quality of life.